CLINICAL TRIAL: NCT04075656
Title: A Pilot Trial of UrApp, a Novel Mobile Application for Childhood Nephrotic Syndrome Management
Brief Title: UrApp for Childhood Nephrotic Syndrome Management (Incident Cohort)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Chia-shi Wang, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00108912; 1K23DK118189-01A1 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Nephrotic Syndrome
Keywords: Pediatrics; mHealth; Behavioral intervention
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UrApp (Experimental): Participants randomized to this study arm will use the UrApp mobile application for one year, in addition to receiving the standard of care.
  Interventions: Behavioral: Standard of Care; Behavioral: UrApp
- Standard of Care (Active Comparator): Participants randomized to this study arm will use receive the standard of care for one year.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Standard of Care — Participants will be provided a folder of educational material on NS, including general information on symptoms, treatments, and possible complications; healthy diet for children taking corticosteroids; and low sodium diet. Site research staff will demonstrate how to check urine for protein with test strips, and educate patients on the definitions of disease relapse and remission. Urine test strips and urine protein logs will be provided to ensure that each participant can check their urine daily for protein. Participants will be instructed to check their urine daily for protein and call their provider within 1 business day for relapses and remissions.
Behavioral: UrApp — Caregivers/parents will download UrApp at the baseline visit. UrApp contains instructional videos to guide users. The telephone number of the patient's provider will be entered into UrApp and participants will be able to call their providers directly through UrApp. The email address of the Emory study staff will also be entered. UrApp will automatically e-mail test results to the research staff when elected by the users. Participants will be asked by study staff, and reminded by the app, to call their providers and send urine testing results to the study staff whenever there is a relapse or remission. When the study staff receives alerts of a relapse/remission via UrApp, the information will be communicated to the treating physician within 1 business day.
  Arms: UrApp

SUMMARY:
Idiopathic nephrotic syndrome is one of the most common chronic kidney diseases in children. Patients suffer from frequent disease relapses and complications. Self-management is difficult for families and nonadherence is common, with adverse effects on the children's health. UrApp is a mobile application designed to assist families with nephrotic syndrome management. This study will examine whether providing the children's caregivers (or adolescent patients) with UrApp improves self-management and disease outcomes. This study will include 60 caregivers of children with newly diagnosed nephrotic syndrome. Participants will be randomized 1:1 to UrApp or standard of care and followed for 1 year.

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome (NS) is one of the most common chronic kidney diseases in children, with a prevalence of approximately 16 cases per 100,000 children. NS is characterized by heavy urinary losses of protein leading to hypoalbuminemia, edema, and hyperlipidemia. Children are treated with high-dose corticosteroids on presentation, and >80% respond to treatment with resolution of proteinuria and symptoms. However, 80-90% of the children initially sensitive to corticosteroids will experience disease relapse, with more than half relapsing frequently or becoming dependent on corticosteroids to maintain remission. During a relapse, patients can suffer from anasarca, acute kidney injury, serious infections, or thromboembolic events.

Management of children with NS entails long-term outpatient surveillance and treatment. Home care includes the important standard-of-care task of urine monitoring to follow the relapsing-remitting nature of the disease. New proteinuria signals disease relapse before the development of overt symptoms such as edema. Thus, patients are instructed to alert their providers to the occurrence of proteinuria in a timely manner so that corticosteroids can be initiated or adjusted to treat each relapse and prevent acute disease complications. It is also important for the patients to track urine protein for resolution so that corticosteroids can be stopped or reduced to minimize steroid toxicity.

Not unlike other chronic, relapsing-remitting pediatric disorders, self-management is difficult for NS patients and their caregivers. Mobile health (mHealth) is a promising, rapidly growing field in disease management. In NS, there are numerous aspects of self-management that may be facilitated by a mobile app. First, the visual analysis of a urine test strip is subject to human error, including reading the wrong reagent block and erroneous assessments of color. This can be improved through using a smartphone's camera and computer to read and analyze test strip results. Second, caregivers must remember to check their child's urine, recall results, and understand what the results mean: the demands are taxing in that disease relapse is defined as urine protein ≥2+ for 3 consecutive days and remission is defined as negative/trace urine protein for 3 consecutive days. Apps, with their inherent interactivity, can provide reminders for urine testing, capture the results, and analyze trends to detect disease relapse/remission. Apps can alert a caregiver to seek medical attention and directly transmit test results to providers. Lastly, apps can provide medication reminders for NS patients, who are on highly complex medication regimens.

UrApp was iteratively developed by an expert panel of two pediatric nephrologists and three research engineers with expertise in human-computer interaction. App features were devised by the clinicians to support elements of chronic care management according to the Chronic Care Model and tasks that are challenging for caregivers. This study will include 60 caregivers of children with newly diagnosed nephrotic syndrome. Participants will be randomized 1:1 to UrApp or standard of care and followed for 1 year. In addition to the study outcome measures, user feedback will be collected via survey, interview, and by stakeholder meetings to inform app refinement.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients ages 1-17 with steroid sensitive nephrotic syndrome (clinical diagnosis with edema, nephrotic range proteinuria [urine protein to creatinine ratio >2 mg/mg, or ≥ 300 mg/dL or ≥ 3+ protein on urine dipstick], and hypoalbuminemia ≤ 2.5 g/dL; resolution of proteinuria [negative/trace protein on urine dipstick] within 4 weeks of corticosteroid treatment)
* Caregivers of pediatric patients with steroid sensitive nephrotic syndrome diagnosed within 42 days at the time of enrollment
* Access to internet/wireless fidelity (Wi-Fi) in the home
* Caregiver proficiency with the English language

Exclusion Criteria:

* Caregivers of pediatric patients with end-stage kidney disease
* Caregivers of pediatric patients with renal transplantation
* Caregivers of pediatric patients with clinical or histologic evidence of secondary nephrotic syndrome (e.g., systemic lupus erythematosus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-shi Wang, MD, MS, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Altanta, Atlanta, Georgia
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available for sharing, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for sharing immediately following publication, with no end date.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to chia-shi.wang@emory.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Derived] Wang CS, Escoffery C, Patzer RE, McCracken C, Ross D, Rheault MN, Al-Uzri A, Greenbaum LA. A dual efficacy-implementation trial of a novel mobile application for childhood nephrotic syndrome management: the UrApp for childhood nephrotic syndrome management pilot study protocol (UrApp pilot study). BMC Nephrol. 2020 Apr 9;21(1):125. doi: 10.1186/s12882-020-01778-w. PMID 32272901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregiver participants were recruited from Children's Healthcare of Atlanta, in Atlanta, Georgia, Oregon Health and Science University, in Portland, Oregon, and the University of Minnesota Children's Hospital in Minneapolis, Minnesota, USA. Participant enrollment began September 17, 2019, and all follow-up assessments were completed by April 25, 2025.
Pre-assignment Details: Caregivers of pediatric patients were enrolled into the study, randomized to a study arm, and took part in the study intervention. Data for outcome measures and adverse events were collected about and from pediatric patients but the study participants are the caregivers rather than pediatric patients.
Groups:
- Caregivers Using UrApp with Standard of Care: Caregiver participants randomized to this study arm use the UrApp mobile application for one year, in addition to receiving the standard of care.
  UrApp: Caregivers/parents download UrApp at the baseline visit. UrApp contains instructional videos to guide users. The telephone number of the patient's provider is entered into UrApp and participants are able to call their providers directly through UrApp. The email address of the Emory study staff is also entered. UrApp automatically e-mails test results to the research staff when elected by the users. Participants are asked by study staff, and reminded by the app, to call their providers and send urine testing results to the study staff whenever there is a relapse or remission. When the study staff receives alerts of a relapse/remission via UrApp, the information is communicated to the treating physician within 1 business day.
- Caregivers Receiving the Standard of Care: Caregiver participants randomized to this study arm receive the standard of care for one year.
  Standard of Care: Participants are provided a folder of educational material on nephrotic syndrome (NS), including general information on symptoms, treatments, and possible complications; healthy diet for children taking corticosteroids; and low sodium diet. Site research staff demonstrate how to check urine for protein with test strips and educate patients on the definitions of disease relapse and remission. Urine test strips and urine protein logs are provided to ensure that each participant can check their urine daily for protein. Participants are instructed to check their urine daily for protein and call their provider within 1 business day for relapses and remissions.
Period: Overall Study
Arm/Group | Caregivers Using UrApp with Standard of Care | Caregivers Receiving the Standard of Care
Started | 30 | 28
Completed (Participants are considered as having completed the study if they contributed any outcome data at either the 6 month or 12 month time points.) | 25 | 23
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- UrApp: Caregiver participants randomized to this study arm use the UrApp mobile application for one year, in addition to receiving the standard of care.
  UrApp: Caregivers/parents download UrApp at the baseline visit. UrApp contains instructional videos to guide users. The telephone number of the patient's provider is entered into UrApp and participants are able to call their providers directly through UrApp. The email address of the Emory study staff is also entered. UrApp automatically e-mails test results to the research staff when elected by the users. Participants are asked by study staff, and reminded by the app, to call their providers and send urine testing results to the study staff whenever there is a relapse or remission. When the study staff receives alerts of a relapse/remission via UrApp, the information is communicated to the treating physician within 1 business day.
- Standard of Care: Caregiver participants randomized to this study arm receive the standard of care for one year.
  Standard of Care: Participants are provided a folder of educational material on nephrotic syndrome (NS), including general information on symptoms, treatments, and possible complications; healthy diet for children taking corticosteroids; and low sodium diet. Site research staff demonstrate how to check urine for protein with test strips and educate patients on the definitions of disease relapse and remission. Urine test strips and urine protein logs are provided to ensure that each participant can check their urine daily for protein. Participants are instructed to check their urine daily for protein and call their provider within 1 business day for relapses and remissions.
- Total: Total of all reporting groups
Arm/Group | UrApp | Standard of Care | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Medication Adherence
Description: Adherence to medications is evaluated via caregiver survey with the validated 4-question Morisky, Green, and Levine (MGL) Adherence Scale. Response options are Yes (0) or No (1) and total scores range from 0 to 4 with higher scores indicating better medication adherence. Adherence will be defined as a score of ≥3 on the MGL scale.
Time Frame: Baseline, Month 6, Month 12
Population: This analysis includes participants who completed the study and responded to this survey. Survey data are missing for some participants. If a participant missed a study visit they were sent the survey electronically but some participants did not complete every survey.
Measure: Count of Participants; unit: Participants
Groups:
- UrApp: Caregiver participants randomized to this study arm use the UrApp mobile application for one year, in addition to receiving the standard of care.
- Standard of Care: Caregiver participants randomized to this study arm receive the standard of care for one year.
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 25 | 22
Participants
  Participants with score ≥3 at Baseline | 25 | 21
  Participants with score ≥3 at Month 6: number analyzed (Participants) | 20 | 19
  Participants with score ≥3 at Month 6 | 19 | 18
  Participants with score ≥3 at Month 12: number analyzed (Participants) | 16 | 18
  Participants with score ≥3 at Month 12 | 15 | 16

2. Primary Outcome: Number of Participants Reporting Adherence With Urine Monitoring
Description: Caregiver adherence with urine protein monitoring is assessed by asking caregivers on average how often they checked their child's urine for protein over the past month. Possible responses are "once a week", "2-4 times a week" or " 5-7 times a week." Adherence is defined as checking urine at least 2 times per week.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 25 | 23
Participants
  Adherence at Baseline | 21 | 18
  Adherence at Month 6: number analyzed (Participants) | 19 | 19
  Adherence at Month 6 | 19 | 18
  Adherence at Month 12: number analyzed (Participants) | 16 | 17
  Adherence at Month 12 | 14 | 14

3. Secondary Outcome: Caregiver Self-efficacy Score
Description: Self-efficacy of caregivers for managing nephrotic syndrome of pediatric patients is assessed with a 3-item instrument adapted from the Chronic Disease Self-Efficacy Scales. Responses are given on a 10-point scale where 0 = not confident at all and 10 = totally confident. Total scores range from 0 to 30 with higher scores indicating increased self-efficacy.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 8.97 (1.84) | 9.35 (1.26)
  Month 6: number analyzed (Participants) | 20 | 19
  Month 6 | 9.65 (1.26) | 9.42 (0.81)
  Month 12: number analyzed (Participants) | 16 | 17
  Month 12 | 9.21 (1.51) | 9.49 (0.88)

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Pediatric Quality of Life Inventory (PedsQL) Score for Parents
Description: The 23-item PedsQL was developed as part of the NIH Roadmap Initiative to create universal measures for patient-reported outcomes and contains questions in the domains of social-peer, depression, anxiety, mobility, and function. Responses are given on a 5-point scale where 0 = never and 4 = almost always. Items are reverse scored and linearly transformed to a scale of 0 to 100, where higher total mean scores indicate a better quality of life.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 25 | 23
score on a scale
  Baseline | 83 (16) | 85 (12)
  Month 6: number analyzed (Participants) | 20 | 19
  Month 6 | 86 (18) | 84 (14)
  Month 12: number analyzed (Participants) | 16 | 17
  Month 12 | 88 (13) | 76 (17)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Pediatric Quality of Life Inventory (PedsQL) Score for Pediatric Patients
Description: The 23-item PedsQL was developed as part of the NIH Roadmap Initiative to create universal measures for patient-reported outcomes, and contains questions in the domains of social-peer, depression, anxiety, mobility, and function. Responses are given on a 5-point scale where 0 = never and 4 = almost always. Items are reverse scored and linearly transformed to a scale of 0 to 100, where higher total mean scores indicate a better quality of life.
Time Frame: Baseline, Month 6, Month 12
Population: This analysis includes pediatric patients who completed the study and responded to this survey. Survey data are missing for some pediatric patients. If a caregiver participant missed a study visit they were sent the survey electronically but some pediatric patients did not complete this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- UrApp: Pediatric patients of caregiver participants randomized to this study arm use the UrApp mobile application for one year, in addition to receiving the standard of care.
- Standard of Care: Pediatric patients of caregiver participants randomized to this study arm receive the standard of care for one year.
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 24 | 23
score on a scale
  Baseline | 91 (7) | 83 (15)
  Month 6: number analyzed (Participants) | 19 | 19
  Month 6 | 89 (10) | 84 (7)
  Month 12: number analyzed (Participants) | 15 | 14
  Month 12 | 94 (5) | 81 (14)

6. Secondary Outcome: Number Pediatric Patients With Delayed Detection of Relapses
Description: Relapses detected only after patients experienced symptoms of relapse, indicating delayed detection, is compared between study arms. Patient medical charts were reviewed for occurrence and frequency of delayed relapse reporting which is defined as a relapse that was not reported to the treating physician until clinical manifestations or complications occurred and/or only discovered during planned or unplanned visits or hospitalizations.
Time Frame: Month 6, Month 12
Population: Information for this outcome measure was collected from medical records. Some participants did not attend clinic visits corresponding with the time frames of this study. The overall number of participants analyzed reflects caregiver participants who contributed data at either the 6 month or 12 month time points, while the number of participants analyzed at each time point are pediatric patients who had a least one relapse during the time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 23 | 22
Participants
  Month 6: number analyzed (Participants) | 18 | 16
  Month 6 | 2 | 7
  Month 12: number analyzed (Participants) | 11 | 14
  Month 12 | 1 | 4

7. Secondary Outcome: Number of Hospitalizations Among Pediatric Patients
Description: Medical records were reviewed for the primary reason for admission and NS disease complications, such as bacterial peritonitis, septicemia, shock, blood clot(s), acute kidney injury, and seizures from hyponatremia or hypertension.
Time Frame: Month 6, Month 12
Population: Information for this outcome measure was collected from medical records. Some participants did not attend clinic visits corresponding with the time frames of this study. The overall number of participants analyzed reflects caregiver participants who contributed data at either the 6 month or 12 month time points, while the number of participants analyzed at each time point are pediatric patients who had medical record data to be reviewed for the indicated study time point.
Measure: Number; unit: count of hospitalizations
Groups:
- UrApp: Pediatric patients of caregiver participants who were randomized to use the UrApp mobile application for one year, in addition to receiving the standard of care.
- Standard of Care: Pediatric patients of caregiver participants who were randomized to receive the standard of care for one year.
Arm/Group | UrApp | Standard of Care
Number analyzed (Participants) | 23 | 20
count of hospitalizations
  Month 6 | 3 | 7
  Month 12: number analyzed (Participants) | 15 | 14
  Month 12 | 4 | 10

ADVERSE EVENTS:
Time Frame: Information on adverse events among pediatric patients was collected beginning one month after initiating the intervention and Months 6 and 12 (up to 11 months).
Description: During study visits, caregivers were asked if their child had any serious illnesses or trips to the hospital since the last study visit. Information on non-serious adverse events among pediatric patients was not collected. Information about adverse events impacting caregiver participants was not collected.
Arm/Group | UrApp | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/30 | 9/28
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UrApp (N=30) | Standard of Care (N=28)
Hospitalization due to anasarca (Renal and urinary disorders) | 4 (4) | 6 (11)
Hospitalization due to fever, concern for infection, or immunosuppression (Infections and infestations) | 3 (3) | 6 (6)
Hospitalization due to peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization due to acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Hospitalization due to electrolyte derangements (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalization due to high blood sugar (Endocrine disorders) | 0 (0) | 1 (1)
Hospitalization due to gastrointestinal parasite (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT04075656/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04075656/ICF_000.pdf